CLINICAL TRIAL: NCT03191461
Title: Myocardial Perfusion and Fibrosis in Cancer Survivors
Status: Completed | Type: Observational
Sponsor: Virginia Commonwealth University (Other)
Collaborators: Wake Forest University (Other)
Responsible Party: Sponsor
Other Study IDs: HM20015409
Record Dates: First submitted 2017-05-25; First posted 2017-06-19 (Actual); Last update posted 2024-10-30 (Actual); Status verified 2024-10

CONDITIONS: Myocardial Fibrosis; Myocardial Injury; Chemotherapeutic Toxicity
Keywords: Anthracycline-based chemotherapy; Anth-bC; Chemotherapy; Myocardial Perfusion
MeSH Terms: interventions — Exercise Test

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

GROUPS / COHORTS (2):
- Cancer Patients: Cancer patients with Stage I-III breast cancer or lymphoma that have received an anthracycline agent during treatment at least 2 years prior to enrollment in this study. Adenosine stress test MRI will be performed.
  Interventions: Diagnostic Test: Adenosine stress test MRI
- Healthy Controls: Age-matched Healthy Control to cancer survivor with no history of cancer or anthracycline treatment. Adenosine stress test MRI will be performed.
  Interventions: Diagnostic Test: Adenosine stress test MRI

INTERVENTIONS:
Diagnostic Test: Adenosine stress test MRI — Participants will receive a contrasted adenosine stress CMR examination on a 1.5T Siemens Avanto scanner (Siemens Medical Solutions, Malvern, PA) dedicated to cardiovascular imaging. Adenosine stress was selected due to attenuated endothelium dependent and -independent vasodilation after doxorubicin receipt in humans to allow the investigators to understand the potential effect of perivascular fibrosis on perfusion reserve. Standardized CMR protocols will be performed to measure LV volumes (to assess wall motion abnormalities and identify any potential myocardial dysfunction), Native T1, ECV, and myocardial perfusion reserve in the short-axis plane
  Other Names: MRI; Stress Test

SUMMARY:
This is a cross-sectional pilot study. The investigators seek to obtain early information pertaining to the relationship between measurements of myocardial perfusion reserve and myocardial fibrosis after receipt of Anthracycline-based chemotherapy (≥2 years prior).

DETAILED DESCRIPTION:
The primary objective of this cross-sectional pilot study is to determine the myocardial perfusion reserve index (MPRI) in cancer survivors treated with anthracycline chemotherapy relative to similarly aged healthy comparators without a history of cancer treatment. Hypothesis: Cancer survivors treated with anthracycline chemotherapy will have a lower MPRI than similarly aged healthy comparators without a history of cancer treatment.The secondary objective of this cross-sectional pilot study is to determine if MPRI is associated with myocardial fibrosis measured non-invasively with cardiovascular magnetic resonance imaging. Hypothesis: MPRI will be inversely associated with fibrosis burden

Study participants will be consented with pre-study data collection recorded. No randomization will occur as this is a cross-sectional study. Participants in both the cancer survivor and control groups will complete one study visit. No follow-up will be completed.

ELIGIBILITY:
Inclusion Criteria :

1. Cancer patients must have Stage I-III breast cancer or lymphoma and have received an anthracycline agent during treatment at least 2 years prior to enrollment in this study.
2. Age-matched to cancer survivor with no history of cancer or anthracycline treatment.
3. Age 21-85 years of age at the time of enrollment.
4. ECOG or Karnofsky performance status of 0-1.
5. Life expectancy of greater than 3 months.
6. Enrolled control participants must have normal creatinine clearance of >60 mL/min/1.73 m2 for patients with creatinine levels above institutional normal.
7. Ability to understand and the willingness to sign an IRB-approved informed consent document (either directly or via a legally authorized representative).

Exclusion Criteria :

1. History of allergic reactions attributed to compounds of similar chemical or biologic composition to gadolinium contrast agents or adenosine or history of kidney disease.
2. Those with contraindications for MRI such as ferromagnetic cerebral aneurysm clips or other intracranial metal, pacemakers, defibrillators, functioning neurostimulator devices or other implanted electronic devices.
3. Uncontrolled intercurrent illness including, but not limited to ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
4. Pregnant women are excluded from this study because the use of gadolinium in cardiac MRI imaging may not be safe in pregnant women. Because some methods of birth control are not 100% reliable, a pregnancy test is required if the participant is a) a sexually active woman of childbearing potential or b) a sexually active peri or post-menopausal women whose last normal menstrual period was less than 12 months ago.
5. Coronary revascularization in the past 6 months or known severe multi-vessel CAD previously determined to be not amendable to mechanical intervention.
6. Ongoing, unrelieved symptoms thought to represent cardiac ischemia and requiring immediate cardiac catheterization
7. History of COPD or asthma

Ages: 21 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The investigators will enroll 10 eligible and consenting men and women aged 21-85 years who either currently have or have had cancer who began their cancer treatment at least 2 years prior to this study and have received anthracycline based chemotherapy. The investigators will enroll an additional group of 6 men and women without cancer or a prior history of a cardiovascular event, matched to 5-year age range with our post-cancer treatment participants
Sampling Method: Non-Probability Sample
Enrollment: 7 (Actual)
Dates: Start 2017-11-13 (Actual); Primary Completion 2024-04-11 (Actual); Study Completion 2024-04-11 (Actual)

PRIMARY OUTCOMES:
Myocardial perfusion reserve index (MPRI) | During Adenosine Stress Test
  The myocardial perfusion reserve index (MPRI) will be measured noninvasively with adenosine stress CMR imaging after dual-bolus first-pass perfusion with gadolinium contrast. The slope of the myocardial signal intensity curve is computed and normalized by the slope of the blood pool signal intensity curve for both rest and stress. MPRI is calculated as the ratio of the stress slope divided by the rest slope.

SECONDARY OUTCOMES:
Myocardial fibrosis quantification using Myocardial T1 | During Adenosine Stress Test
  Measured noninvasively with CMR imaging. For myocardial fibrosis quantification with T1 endocardial and epicardial contours are drawn to delineate the myocardium; mean T1 (pre- and post-contrast) is calculated from the pixels within the myocardium. Expected range of T1 is 900-1250ms with higher T1 values considered a worsened outcome.
Myocardial fibrosis quantification using extracellular volume (ECV) | During Adenosine Stress Test
  Measured noninvasively with CMR imaging. The ECV is calculated from the mean myocardial T1 and LV blood T1 pre- and post-contrast. Expected range of ECV is 20-40% with higher ECV values representing a worse outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer H Jordan, PhD, Principal Investigator — Virginia Commonwealth University
Locations (2):
- United States (2):
  - Wake Forest Baptist Heath, Winston-Salem, North Carolina
  - Virginia Commonwealth University, Richmond, Virginia

IPD SHARING:
Plan to Share IPD: No